CLINICAL TRIAL: NCT01287611
Title: Short Term Comparison of Double Layer Continuously Locked Closure of Uterine Incision in Cesarean Section Versus Double Layer Purse String Closure (Turan Technique): A Prospective Randomized Study
Brief Title: Short Term Comparison of Two Different Techniques of Uterine Cesarean Incision Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Cem Turan, Chief Clinical, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kartal1; 21.01.2011-02(1) (Other: Ethics committee ID number)
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean section; Kerr incision; Purse string suturing in C/S; Continuous locked suturing in C/S

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purse string closure technique (Active Comparator): Eighty four patients were allocated to the study group. Due to expanded Kerr incisions 4 patients in study group did not receive their allocated intervention. In addition, 29 patients in the study group were lost to follow up and did not come to the sixth week check up. Statistical analysis is based on data from the remaining 51 study group.
  Interventions: Procedure: Purse string closure technique
- Continuously locked closure technique (Active Comparator): Eighty four patients were allocated to the control group. Due to expanded Kerr incisions 3 patients in control group did not receive their allocated intervention. In addition, 16 patients in the control group were lost to follow up and did not come to the sixth week check up. Statistical analysis is based on data from the remaining 65 study group.
  Interventions: Procedure: Continuously locked closure technique

INTERVENTIONS:
Procedure: Purse string closure technique — Uterine Kerr incision will be closed with purse string suture
  Other Names: Uterine incision in C/S
  Arms: Purse string closure technique
Procedure: Continuously locked closure technique — Uterine Kerr incision will be closed with continuously locked suturing
  Other Names: Uterine incision in C/S
  Arms: Continuously locked closure technique

SUMMARY:
Cesarean section (C/S) is an operation most commonly performed in Obstetrics and Gynecology Clinics. Complications related with incomplete healing of Kerr uterine incision after C/S (adhesions, separation (dehiscence), endometritis, endometriosis, anomalous placentation in subsequent pregnancies, incomplete or complete uterine rupture in subsequent pregnancies, ...) are very important issues. Classically Kerr incision is repaired with continuous locked suturing. Purse string suturing of Kerr incision may reduce the size of the incision and in turn may reduce short and long term complications. For this reason, the investigators aimed to compare two closure techniques.

DETAILED DESCRIPTION:
In the clinic, patients undergoing cesarean section that meet the criteria for inclusion into the study and agreed to participate in the study will be randomized into two groups (computer-assisted randomization method will be used.) In the first group of patients classical closure method of Kerr incision (double layered continuously locked suturing) will be used. In the second group of patients double layered purse string closure technique will be used. The two groups will be compared after 6 weeks in terms of healing, operation time, blood loss, incision size and incisional scar defect( if present). A physician who does not know the method of closure will evaluate incision size by transabdominal and/or transvaginal ultrasound. The length of the incision and myometrial thickness in Kerr incisional line will be measured and recorded in longitudinal and transverse axis separately. If any incisional scar defect is determined it will be measured and recorded also.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term (> 37 weeks) pregnancy
* Cervical dilatation < 4 cm
* Kerr incision
* Age > 18 years old

Exclusion Criteria:

* Being in active phase of labor
* Emergency situations (fetal distress, cord prolapse, placental abruption,severe pre-eclampsia, eclampsia, placenta previa, vasa previa )
* Having a history of uterine surgery (myomectomy, hysterotomy)other than C/S
* Extension of Kerr incision
* Multiple pregnancy
* Maternal diabetes mellitus
* Maternal connective tissue disease
* Uterine malformation
* Uterine fibroids on Kerr incision line
* Chorioamnionitis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Karsidağ, Study Chair — Dr. Lutfi Kirdar Kartal Education and Research Hospital
Locations (1):
- Dr. Lütfi Kirdar Kartal Education and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

REFERENCES:
- [Background] Turan C, Buyukbayrak EE, Yilmaz AO, Karsidag YK, Pirimoglu M. Purse-string double-layer closure: a novel technique for repairing the uterine incision during cesarean section. J Obstet Gynaecol Res. 2015 Apr;41(4):565-74. doi: 10.1111/jog.12593. Epub 2014 Nov 5. PMID 25370526
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov/25370526/
- See also: The video of purse string uterine closure (Turan Technique) in cesarean section — http://www.dailymotion.com/video/x2fxlgp_closure-of-uterine-incision-in-cesarean-section-with-turan-technique_school

RESULTS

PARTICIPANT FLOW:
Groups:
- Purse String Closure Technique: Purse string closure: Uterine Kerr incision will be closed with purse string suture
- Continuously Locked Closure Technique: Continuously locked suturing: Uterine Kerr incision will be closed with continuously locked suturing
Period: Overall Study
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Started | 84 | 84
The Number of Patients Who Underwent C/S | 84 | 84
Completed | 51 | 65
Not Completed | 33 | 19
Not completed — Lost to Follow-up | 29 | 16
Not completed — Exclusion due to expanded Kerr incision | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique | Total
Number analyzed (Participants) | 51 | 65 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.0) | 28.5 (5.3) | 29.05 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 65 | 116
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 51 | 65 | 116

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Scar Defect in the Uterine Incisional Line
Description: A wedge-shaped distortion in the integrity of the uterine incision scar during transvaginal ultrasonographic examination at 6 weeks after C/S was accepted as cesarean scar defect in the uterine incisional line and recorded as primary outcome measure, and two groups will be compared.
Time Frame: 6 weeks after C/S
Measure: Number; unit: participants
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 51 | 65
participants | 12 (4.38) | 39 (6.11)
Statistical Analysis 1: Comparison: Purse String Closure Technique vs Continuously Locked Closure Technique; Test type: Non-Inferiority or Equivalence — Group sample sizes of 51 in study group and 65 in control group achieve 98% power to detect a difference between the group proportions of -0.3300. The proportion in study group is assumed to be 0.4800 under the null hypothesis and 0.1500 under the alternative hypothesis. The proportion in control group is 0.4800. The test statistic used is the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.0500; p = 0.0001, Chi-squared

2. Secondary Outcome: Length of Uterine Incision After Suturing
Description: Length of uterine incision after suturing will be examined and measured by ultrasonography, and two groups will be compared.
Time Frame: 6 weeks after C/S
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 51 | 65
cm | 3.7 (0.9) | 8.5 (1.7)
Statistical Analysis 1: Comparison: Purse String Closure Technique vs Continuously Locked Closure Technique; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/65
Other Adverse Events (participants affected / at risk) | 0/51 | 0/65

LIMITATIONS AND CAVEATS:
The present trial is a single-center study. The similar results should be supported in a multicenter study. Another limitation of this study is the more than 25% overall rate of loss to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No